CLINICAL TRIAL: NCT07375290
Title: Early Intervention With Zoledronate to Safely Prevent Bone Health Complications in Pediatric Hematopoietic Stem Cell Transplant Survivors
Brief Title: Zoledronate to Prevent Bone Health Complications in Pediatric Hematopoietic Stem Cell Transplant Survivors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0052
Record Dates: First submitted 2025-11-12; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Zoledronate (Experimental): Zoledronate dose will be given intravenously over 1 hour using standard infusion equipment. Patients will receive a dose of 0.025 mg/kg. Zoledronate will be infused in the inpatient setting to facilitate proper observation and data collection.
  Interventions: Drug: Zoledronate

INTERVENTIONS:
Drug: Zoledronate — Zoledronate is in the class of drugs entitled bisphosphonates which act to inhibit bone resorption by inhibiting osteoclast activity therefore reducing bone turnover.

SUMMARY:
The purpose of this pilot study is to investigate the safety and preliminarily assess efficacy of early intervention with zoledronate in high risk pediatric hematopoietic stem cell transplantation (HSCT) patients to prevent the development of bone disease and fractures and reduce potential pain and suffering.

DETAILED DESCRIPTION:
Bone disease, including low bone density and fragility fractures (osteoporosis), is common among survivors of pediatric hematopoietic stem cell transplantation (HSCT). Further, patients who develop graft-versus-host disease (GVHD) following HSCT or who have high cumulative doses of glucocorticoids are at even higher risk to develop bone complications. Recent data also suggest that a large number of HSCT candidates arrive to transplantation already with low bone mineral density, adding to the potential risk of developing bone disease following HSCT. Typically, treatment for osteoporosis in children using bisphosphonates, such as zoledronate, is recommended only after the development of fragility fractures.

The investigators propose to study the safety and efficacy of a novel method of early intervention with zoledronate in high risk pediatric HSCT patients to prevent the development of bone disease and fractures in order to reduce potential pain and suffering.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥5 and ≤18 years old who are preparing for HSCT with a height-for-age corrected DXA Z-score of <-2.0 and admitted to a CCHMC inpatient unit.
* Patients ≥5 and ≤18 years old recovering from HSCT and who have developed de novo acute or chronic GVHD and are admitted to a CCHMC inpatient unit.

Exclusion Criteria:

* Age <5 years and >18 years
* Patients with Fanconi anemia or other radiation-sensitive syndromes with increased malignancy risk
* history of prior bisphosphonate use
* low 25-OH vitamin D levels (<20 ng/mL)
* active febrile illness
* uncontrolled infection
* Elevated creatinine at the time of enrollment, history or renal failure, or documented low glomerular filtration rate (GFR≤90)
* Active bone disease including history of abnormal PTH level for any reason, active bone fracture/healing, or primary disorder of bone development or metabolism.
* Women who are pregnant or breast feeding.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Safety of early intervention Zoledronate | At the time of infusion through up to 60 days post last dose of Zoledronate
  Calcium levels following infusion of zoledronate
Feasibility of early intervention Zoledronate | At patient discharge, typically 1 week post infusion
  Number of days required for inpatient stay beyond what is necessary for the patient's admission

SECONDARY OUTCOMES:
Bone health efficiency | Baseline, +6 months, and +12 months
  DXA scans will be measured with a z-score comparing bone density to averages for patient age and height
Bone substrate turnover | Baseline and +30 days
  c-terminal telopeptide (CTX) and procollagen type 1 n-terminal propeptide (P1NP) measured in pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No